CLINICAL TRIAL: NCT02276209
Title: A Randomized, Double Blind, Multicenter, Placebo Controlled, Parallel Group, Efficacy and Safety Study of 2 Doses of Dasotraline in Adults With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: Dasotraline Adult ADHD Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Sumitomo Pharma America, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SEP360-301
Record Dates: First submitted 2014-10-21; First posted 2014-10-28 (Estimated); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Adult Attention Deficit Hyperactivity Disorder
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity | interventions — 4-(3,4-dichlorophenyl)-1,2,3,4-tetrahydronaphthalen-1-amine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Dasotraline 4 mg (Experimental): Dasotraline 4 mg once daily
  Interventions: Drug: Dasotraline
- Dasotraline 6 mg (Experimental): Dasotraline 6 mg once daily
  Interventions: Drug: Dasotraline
- Placebo (Placebo Comparator): Placebo once daily
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Dasotraline — Dasotraline 4 mg once daily
  Arms: Dasotraline 4 mg
Drug: Dasotraline — Dasotraline 6 mg once daily
  Arms: Dasotraline 6 mg
Other: Placebo — Placebo once daily
  Arms: Placebo

SUMMARY:
This is a randomized, double blind, multicenter, parallel group, outpatient study evaluating the efficacy and safety of dasotraline in adults with ADHD.

DETAILED DESCRIPTION:
This is a randomized, double blind, multicenter, parallel group, outpatient study evaluating the efficacy and safety of dasotraline in adults with ADHD using 2 doses of dasotraline (4 mg/day or 6 mg/day) versus placebo over an 8 week treatment period (8 weeks of active treatment followed by a 2-week withdrawal phase).

ELIGIBILITY:
Inclusion Criteria:

* Subject is male or female, 18 to 55 years old, inclusive, at the time of informed consent.
* Diagnostic and Statistical Manual of Mental Disorders Fifth Edition (DSM 5) criteria for a primary diagnosis of ADHD (inattentive, hyperactive, or combined subtype) established by a comprehensive psychiatric evaluation that reviews psychiatric criteria. Diagnosis is confirmed by Adult ADHD Clinical Diagnostic Scale (ACDS). Note: The diagnosis of ADHD and appropriateness of inclusion in the trial will be independently confirmed by external expert review. Experts will review diagnostic and other screening instruments for each subject and approval is required before a subject can be randomized. The Mini International Neuropsychiatric Interview (MINI) will be administered to confirm the absence of any other comorbid psychiatric disorders.
* Subject has an ADHD RS IV with adult prompts total score of ≥ 26 at screening and at Baseline.
* Subject has a CGI S score of ≥ 4 at screening and at Baseline.
* Subject has a negative breath alcohol test and a negative urine drug screen (UDS) for any illicit drug at screening.
* If the subject has a positive drug screen for ADHD medications (eg, amphetamine) at screening, the subject must have a negative repeat UDS at least 7 days before baseline.
* Subject is male or a non pregnant, non lactating female.
* Female subjects must have a negative serum pregnancy test at screening; females who are post menopausal (defined as at least 12 months of spontaneous amenorrhea) and those who have undergone hysterectomy or bilateral oophorectomy will be exempted from the pregnancy test.
* Female subjects of childbearing potential and male subjects with female partners of childbearing potential must agree to use an effective and medically acceptable form of birth control, as defined in Section 10.4, throughout the study period. Note: Continued use of an effective and medically acceptable form of birth control is recommended for 30 days after study completion.
* Subject must have a stable living arrangement that allows for consistent participation for the full duration of the study.
* Subject must be able to comply with study medication administration and adhere to protocol requirements.
* Subject can read well enough to understand the informed consent form and other subject materials.
* Subjects must complete a practice trial for the TASS assessment at one timepoint during Screening.

Exclusion Criteria:

* Subject has a ≥ 25% improvement on the ADHD RS IV total score between screening and baseline.
* Subject has a psychiatric disorder other than ADHD that has been the primary focus of treatment at any time during the 12 months before screening.
* Subject has a past history of, or current presentation consistent with, bipolar disorder (including bipolar I and bipolar II), schizophrenia, schizoaffective disorder, or any other psychotic disorder; a personality disorder per DSM 5 criteria.
* Subject has a history of drug dependence or Substance Related Disorder (excluding nicotine and caffeine) within the 12 months before screening, as defined by DSM 5 criteria.

  -- Subject has Hamilton Anxiety Rating Scale (HAM A) total score ≥ 21 at screening and baseline.
* Subject has PSQI total score ≥ 8 at screening or baseline or moderate to severe insomnia as determined by the Investigator.
* Subject has a history of non-response (per clinician judgment) to two adequate treatment regimens of stimulant or non-stimulant treatment for ADHD.
* Subject has a history of epilepsy, seizures (except childhood febrile seizures), unexplained syncope or other unexplained blackouts (except single incident), or head trauma with loss of consciousness lasting more than 5 minutes, or a history of clinically significant multiple head traumas without loss of consciousness.
* Subject has an acute or chronic medical condition (other than ADHD) that in the opinion of the investigator could confound clinical assessments or interfere with the ability of the subject to participate in the study.
* Subject is currently taking or has taken within 6 weeks prior to screening an antidepressent medication; antipsychotic medication; or lithium (any lithium preparation or formulation).
* Subject is currently taking or has taken within the previous 6 months an anticonvulsant medication (eg, phenytoin, carbamazepine, lamotrigine, valproic acid); antipsychotic medication; or lithium (any lithium preparation or formulation).
* Subject is currently taking an alpha 2 adrenergic receptor agonist (including clonidine and guanfacine).
* Subject has a life-time history of a pattern of abuse or diversion of stimulants.
* Subject has a body mass index (BMI) less than 18 or greater than 35 kg/m2 at screening or baseline.
* Subject answers "yes" to "suicidal ideation" item 4 (active suicidal ideation with some intent to act, without specific plan) or item 5 (active suicidal ideation with specific plan and intent) on the C SSRS assessment at screening (in the past month). Subjects who answer "yes" to this question must be referred to the Investigator for follow up evaluation.
* Subject has attempted suicide within 2 years before the screening period.
* Subject has history of positive test for Hepatitis B surface antigen or Hepatitis C antibody and has liver function test results at screening above the upper limit of normal (ULN) for the reference laboratory.
* Subject is known to have tested positive for human immunodeficiency virus (HIV).
* Subject has a clinically significant abnormality on screening evaluation including physical examination, vital signs, ECG, or laboratory tests that the Investigator considers to be inappropriate to allow participation in the study.
* The subject's screening ECG shows a corrected QT interval using Fridericia's formula (QTcF) of ≥ 450 msec for male subjects or ≥ 470 msec for female subjects. Eligibility will be based on the core laboratory ECG interpretation report.
* The subject's screening hematology results show an alanine aminotransferase (ALT) or aspartate aminotransferase (AST) value ≥ 2 times the ULN, or a blood urea nitrogen (BUN) value ≥ 1.5 times the ULN for the reference range.
* Subject has a history of allergic reaction or has a known or suspected sensitivity to any substance that is contained in the study medication formulation.
* Subject is currently participating or has participated in a clinical trial within the last 90 days or has participated in more than 2 clinical trials within the past year. This includes studies using marketed compounds or devices. Note: Subjects will be checked for multiple study enrollments by site staff.
* Subject has been incarcerated in a prison within 12 months prior to Screening.
* Subject has previously been randomized in a clinical trial of dasotraline.
* Subject is an investigational site staff member or the relative of an investigational site staff member.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 636 (Actual)
Dates: Start 2014-12; Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Change from baseline at Week 8 in ADHD symptoms measured by the ADHD Rating Scale Version IV (ADHD RS IV) with adult prompts total score. | 8 Weeks

SECONDARY OUTCOMES:
Change from baseline in ADHD symptoms measured with the ADHD Rating Scale Version IV (ADHD RS IV) with adult prompts total score at Weeks 1, 2, 4, and 6. | 8 Weeks
Change from baseline in the inattentiveness and hyperactivity-impulsivity subscale scores of the ADHD Rating Scale Version IV (ADHD RS IV) with adult prompts at Weeks 1, 2, 4, 6, and 8. | 8 Weeks
Change from baseline in Clinical Global Impression - Severity scale (CGI S) scale at Weeks 1, 2, 4, 6, and 8. | 8 Weeks
Change from baseline in Sheehan Depression Scale (SDS) total score at Weeks 4 and 8. | 8 Weeks
Change from baseline in Sheehan Depression Scale (SDS) domain scores: work/school, family life, social life at Weeks 4 and 8. | 8 Weeks
Change from baseline in Behavior Rating Inventory of Executive Function®-Adult Version (BRIEF A) Global Executive Composite score and Behavioral Regulation Index (BRI) and Metacognition Index (MI) at Weeks 4 and 8. | 8 Weeks
Change from baseline in ADHD Impact Module - Adult AIM A in global domain scores at Weeks 4 and 8. | 8 Weeks
Time sensitive ADHD Symptom Scale (TASS) total score and subscale scores (Inattention and Hyperactive impulsive) at Weeks 3, 5, and 7. | 8 Weeks
Change from baseline in Adult ADHD Self Report Scale (Version 1.1) (ASRS) total score and subscale scores (inattention, hyperactivity-impulsivity, executive function, emotional control, and impulsivity) at each week. | 8 Weeks
Adult ADHD Medication Smoothness of Effect Scale (AMSES) score at Weeks 2, 4, 6, and 8. | 8 Weeks
Change from baseline in Pittsburgh Sleep Quality Index (PSQI) global score and 7 component scores at Weeks 2, 4, and 8. | 8 Weeks
The incidence of overall AEs, serious AEs (SAEs), and AEs (or SAEs) leading to discontinuations. | 8 Weeks
Clinical laboratory evaluations (serum chemistry). | 8 Weeks
Clinical laboratory evaluations ( lipid panel). | 8 Weeks
Clinical laboratory evaluations (thyroid function panel). | 8 Weeks
Clinical laboratory evaluations (hematology). | 8 Weeks
Clinical laboratory evaluations (urinalysis). | 8 Weeks
Clinical evaluations (vital signs). | 8 Weeks
Clinical evaluations (orthostatic effects). | 8 Weeks
Clinical evaluations (physical examinations). | 8 Weeks
Clinical evaluations (body weight). | 8 Weeks
Clinical evaluations (12 lead ECGs). | 8 Weeks
Frequency and severity of suicidal ideation and suicidal behavior as assessed by the C SSRS. | 8 Weeks
Drug Effects Questionnaire (DEQ) scores at Weeks 1, 2, 4, 6, and 8. | 8 Weeks
Symptoms of withdrawal by Physician Withdrawal Checklist (PWC) scores at Week 8, 9, and 10. | 10 Weeks
Symptoms of withdrawal by Study Medication Withdrawal Questionnaire (SMWQ) scores at Weeks 9 and 10. | 10 Weeks
Symptoms of withdrawal by Hamilton Anxiety Rating Scale (HAM A) scores at Weeks 8, 9, and 10. | 10 Weeks
Symptoms of withdrawal by Montgomery-Asberg Depression Rating Scale (MADRS) scores at Weeks 8, 9, and 10. | 10 Weeks

CONTACTS AND LOCATIONS:
Overall Officials: SEP-289 Medical Director, MD, Study Director — Sumitomo Pharma America, Inc.
Locations (59):
- United States (59):
  - NoesisPharma,LLC, Phoenix, Arizona
  - Preferred Research Partners, Little Rock, Arkansas
  - Southern California Research LLC, Beverly Hills, California
  - Pharmacology Research Institute, Encino, California
  - Collaborative Neuroscience Network, LLC, Garden Grove, California
  - North County Clinical Research, Oceanside, California
  - University ot California, San Francisco, San Francisco, California
  - Elite Clinical Trials, Inc., Wildomar, California
  - MCB Clinical Research Centers, LLC, Colorado Springs, Colorado
  - ConnecticutClinicalResearch, Cromwell, Connecticut
  - CNS Clinical Research Group, Coral Springs, Florida
  - Gulfcoast Clinical Research, Fort Myers, Florida
  - Clinical Neuroscience Solutions, Inc., Jacksonville, Florida
  - Florida Clinical Research Center, LLC, Maitland, Florida
  - Miami Research Associates, Miami, Florida
  - Clinical Neuroscience Solutions, Inc., Orlando, Florida
  - Meridien Research, Tampa, Florida
  - The Institute for Advanced Medical Research, Alpharetta, Georgia
  - Atlanta Center for Medical Research, Atlanta, Georgia
  - iResearch Atlanta, LLC, Decatur, Georgia
  - Northwest Behavioral Research Center, Roswell, Georgia
  - Carman Research, Smyrna, Georgia
  - Capstone Clinical Research, Inc., Libertyville, Illinois
  - Alpine Clinic, Lafayette, Indiana
  - Lake Charles Clinical Trials, Lake Charles, Louisiana
  - Kennedy Krieger Institute, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - Neurobehavioral Medicine Group, Bloomfield Hills, Michigan
  - Rochester Center for Behavioral Medicine, Rochester Hills, Michigan
  - Saint Charles Psychiatric Associates/Midwest Research Group, Saint Charles, Missouri
  - Midwest Research Group, Saint Charles, Missouri
  - Premier Psychiatric Research Institute, LLC, Lincoln, Nebraska
  - Center for Emotional Fitness, Cherry Hill, New Jersey
  - Village Clinical Research Inc., New York, New York
  - NYU School of Medicine, New York, New York
  - Eastside Comprehensive Medical Center, LLC, New York, New York
  - Finger Lakes Clinical Research, Rochester, New York
  - Duke Child and Family Study Center, Durham, North Carolina
  - Triangle Neuropsychiatry, Durham, North Carolina
  - University of Cincinnati, Department of Psychiatry, Cincinnati, Ohio
  - IPS Research Company, Oklahoma City, Oklahoma
  - Paradigm Research Professionals, Oklahoma City, Oklahoma
  - SummitResearchNetwork, Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Portland, Oregon
  - Oregon Center for Clinical Investigations, Inc., Salem, Oregon
  - Keystone Clinical Studies, LLC, Norristown, Pennsylvania
  - Medical University of SC (MUSC), Charleston, South Carolina
  - Coastal Carolina Research Center, Mt. Pleasant, South Carolina
  - FutureSearch Clinical Trials, LP, Austin, Texas
  - FutureSearch Trials of Dallas, LP, Dallas, Texas
  - Pillar Clinical Research, LLC, Dallas, Texas
  - Bayou City Research Corporation, Houston, Texas
  - Clinical Trials of Texas, Inc, San Antonio, Texas
  - Road Runner Research, San Antonio, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Neuropsychiatric Associates, Woodstock, Vermont
  - NeuroScience, Inc, Herndon, Virginia
  - Summit Research Network LLC, Seattle, Washington
  - Dean Foundation for Health, Research and Education, Middleton, Wisconsin

REFERENCES:
- [Derived] Adler LA, Goldman R, Hopkins SC, Koblan KS, Kent J, Hsu J, Loebel A. Dasotraline in adults with attention deficit hyperactivity disorder: a placebo-controlled, fixed-dose trial. Int Clin Psychopharmacol. 2021 May 1;36(3):117-125. doi: 10.1097/YIC.0000000000000333. PMID 33724251